CLINICAL TRIAL: NCT03384433
Title: Safety and Efficacy of Allogenic Mesenchymal Stem Cells Derived Exosome on Disability of Patients With Acute Ischemic Stroke: a Randomized, Single-blind, Placebo-controlled, Phase 1, 2 Trial
Brief Title: Allogenic Mesenchymal Stem Cell Derived Exosome in Patients With Acute Ischemic Stroke
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: Tarbiat Modarres University (Other)
Responsible Party: Principal Investigator, Leila Dehghani, Dr Masoud Soleimani, Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: med shahid beheshti university
Record Dates: First submitted 2017-11-29; First posted 2017-12-27 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Cerebrovascular Disorders
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- exosome or vesicle (Experimental): CVA patients who have disability, will receive total protein of allogenic MSC-generated exosome transfected by miR-124, one month after attack, via Stereotaxis/Intraparanchymal
  Interventions: Biological: exosome

INTERVENTIONS:
Biological: exosome — allogenic mesenchymal stem cells derived exosome enriched by miR-124

SUMMARY:
Administration of cell-free exosomes derived from mesenchymal stem cell (MSCs) can be sufficient to exert therapeutic effects of intact MSCs after brain injury. In this study we aim to assay the administration of MSC derived exosome on improvement of disability of patients with acute ischemic stroke

DETAILED DESCRIPTION:
Exosomes derived from multipotent mesenchymal stromal cells (MSCs) promote neurovascular remodeling and functional recovery after stroke. Animal study has shown that Exosome treatment markedly increased the number of newly formed doublecortin (a marker of neuroblasts) and von Willebrand factor (a marker of endothelial cells) cells. Based on previous literature, intravenous administration of MSC-generated exosomes post stroke improves functional recovery and enhances neurite remodeling, neurogenesis, and angiogenesis and represents a novel treatment for stroke. Also some studies have presented which miR-124-Loaded Exosomes ameliorate the brain Injury by promoting neurogenesis. So in present study we aim to assess improving patients with acute ischemic stroke who received MSC derived exosome

ELIGIBILITY:
Inclusion Criteria:

* Male or female acute ischemic patients aged 40-80 years with symptoms of acute cerebral infarction of less than 24h from stroke onset.
* Patients with infarct size 3*3
* Patients with a measurable focal neurological that must persist to the time of treatment without clinically meaningful improvement.
* Patients must have computerized tomography (CT) and / or magnetic resonance imaging (MRI) compatible with the clinical diagnosis of acute ischemic stroke in the territory of the middle cerebral artery before being included in the study.
* Patients must have a score on the NIH Stroke Scale 8-24, and mRS ≤ 1
* Women of childbearing age should have a negative pregnancy test performed prior to inclusion
* Obtaining informed consent signed

Exclusion Criteria:

Comatose patients.

* brain tumour, cerebral oedema with compression of ventricles, cerebellar infarction or brainstem, or intraventricular, intracerebral or subarachnoid haemorrhage.
* alcohol use Active infectious disease, including HIV, hepatitis B, Hepatitis .
* patients with dementia.
* Specify clinical conditions
* Patients who are participating in another clinical trial.
* Inability or unwillingness of individual for giving written informed consent.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2021-06-17 (Estimated); Study Completion 2021-12-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 months
  deteriorating stroke, stroke recurrences, brain oedema, seizures, hemorrhagic transformation

SECONDARY OUTCOMES:
measurement of Modified Ranking Scale | 12 months
  measure the degree of disability in Stroke patients. score was recorded from 0-6.
  0 No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead

CONTACTS AND LOCATIONS:
Overall Officials: Saeed Oraee-Yazdani, Dr, Study Director — Shahid Beheshti University of Medical Sciences
Locations (1):
- Shahid Beheshti University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aldali F, Deng C, Nie M, Chen H. Advances in therapies using mesenchymal stem cells and their exosomes for treatment of peripheral nerve injury: state of the art and future perspectives. Neural Regen Res. 2025 Nov 1;20(11):3151-3171. doi: 10.4103/NRR.NRR-D-24-00235. Epub 2024 Oct 22. PMID 39435603